CLINICAL TRIAL: NCT02179593
Title: Effectiveness of Surgically Assisted Rapid Palatal Expansion (SARPE) With 3 and 2-Segment Technique: A Randomized Clinical Trial
Brief Title: Effectiveness of SARPE With 3 and 2-Segment Technique: A Randomized Clinical Trial
Acronym: 3S/2S_SARPE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Federal University of São Paulo (Other)
Responsible Party: Principal Investigator, Max Domingues Pereira, MD, PhD, Federal University of São Paulo
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: 464.869
Record Dates: First submitted 2014-06-29; First posted 2014-07-02 (Estimated); Last update posted 2016-03-16 (Estimated); Status verified 2016-03

CONDITIONS: Maxillary Hypoplasia
Keywords: Maxillary expansion; Orthognathic surgery; Symmetry; Palatal expansion technique; Maxilla abnormality
MeSH Terms: conditions — Retrognathia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 2-Segment SARPE (Other): Maxilla expansion using one sagittal section of the maxilla.
  Interventions: Other: 2-Segment SARPE
- 3-Segment SARPE (Other): Maxilla Expansion using two parasagittal section of the maxilla.
  Interventions: Other: 3-Segment SARPE

INTERVENTIONS:
Other: 2-Segment SARPE — Le Fort I osteotomy with oppening of the median palatal suture and SARPE.
  Other Names: Surgically Assisted Rapid Maxillary Expansion (SARME); Surgically Assisted Rapid Palatal Expansion (SARPE)
  Arms: 2-Segment SARPE
Other: 3-Segment SARPE — Le Fort I osteotomy with two parallel osteotomies symetrically positioned with reference to the median palatal suture and SARPE.
  Other Names: Surgically Assisted Rapid Palatal Expansion (SARPE); Surgically Assisted Rapid MaxillaryExpansion (SARME)
  Arms: 3-Segment SARPE

SUMMARY:
A few studies state that 3-segment SARPE has the following advantages: a) higher level of expansion symmetry; b) higher level of stability of the expansion achieved; and c) faster bone healing. The investigators hypothesize that 2-segment SARPE is as effective as 3-segment SARPE concerning treatment and/or quality of life in daily practice.

DETAILED DESCRIPTION:
32 healthy, literate adult patients (male and female) with 7-millimeter transverse maxilla deficiency bilaterally distributed will participate in this study.

The participants will be assigned randomizable in equal number to undergo either 3-segment or 2-segment SARPE.

Individuals that a) have undergone maxilla surgery previously; b) have craniofacial anomaly;and c) have dental crowding will not be enrolled.

All participants will be assessed before and after surgery for sensitivity to pressure and temperature in the innervated structures linked to the maxilla, as well as for quality of life using OHIP-49 and B-OQLQ assessment tools.

The expansion of maxilla will be assessed by superimposing tomographic images before and after surgery.

ELIGIBILITY:
Inclusion Criteria:

* Being healthy and literate
* Having 7-millimeter transverse maxilla deficiency bilaterally distributed.

Exclusion Criteria:

* Having undergone maxilla surgery previously
* Having craniofacial anomaly
* Having excessive dental crowding.

Ages: 17 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 50 (Estimated)
Dates: Start 2013-09; Primary Completion 2016-08 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Quality of Life | An average of 2 weeks after expansion.
  The primary outcome chosen in this study is Quality of Life assessed through the Orthognathic Quality of Life Questionaire (OQLQ) and Oral Health Impact Profile (OHIP-49) currently available in Portuguese language and validated for scientific studies.

SECONDARY OUTCOMES:
Maxillary symmetry | pre-operative and an average of 2 weeks at the end of maxillary expansion.
  The maxillary symmetry will be assessed by analyzing before and after 3D imaging obtained from computed tomography data , superimposed using the Geomagic Qualify software.
Stability of dental and osseous structures | pre-operative, an average of 2 weeks at the end of the expansion, 4 months, 1 and 2 years after maxillary expansion.
  The stability of dental and osseous structures will be analyzed using computer-aided 3D analysis of data obtained through the scanning of dental casts using Bicam 3D scanner (Scaierman - Italy).
Nasal and paranasal topographic changes | pre-operative,an average of 2 weeks at the end of the expansion, 4 and 12 months after maxillary expansion.
  The nasal and paranasal topographic changes will be captured using laser scanner device.

CONTACTS AND LOCATIONS:
Overall Officials: Max D Pereira, PhD, Principal Investigator — Federal University of São Paulo; Gabriela PR Prado, MS, Study Chair — Federal University of São Paulo; Fabianne MG Furtado, PhD, Study Chair — Federal University of São Paulo; Lydia M Ferreira, PhD, Study Chair — Federal University of São Paulo
Locations (1):
- Federal University of Sao Paulo, São Paulo, São Paulo, Brazil